CLINICAL TRIAL: NCT00825461
Title: Level of Ghrelin With Anorexia Nervosa (AN) Patients. Subgroup AN: With and Without Tubefeeding.
Brief Title: Ghrelin With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-3-089
Record Dates: First submitted 2009-01-20; First posted 2009-01-21 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2009-09

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- 1: Anorexia with tube feeding
- 2: Anorexia without tube feeding
- 3: Control

SUMMARY:
The PICOWO research group in corporation with the University of Amsterdam (Artificial Intelligence) has developed a computer simulationmodel of eating disorders (Bosse, Delfos, Jonker & Treur, 2003). In a running Phd project we want to add ghrelin to the model. The idea for this current research is to collect clinical information about the functioning and (patho)physiology of ghrelin in patients with AN, so we can extend the simulation.

DETAILED DESCRIPTION:
Eating disorders are in need of new perspectives. A better understanding of the appetite in patients with eating disorders, especially Anorexia Nervosa, could be investigated by the levels of ghrelin in patients with and without tube feeding.

ELIGIBILITY:
Inclusion Criteria:

* Studypopulation: Patiënts: all female, non -age coupled.
* Subgroup patients without tube feeding, with tube feeding and a healthy matched control group.
* Control group: healty volunteers of the University of Maastricht.

Exclusion Criteria:

* Patients with a history of eating disorder different than AN or a psychiatric history.
* Control group: no history of eating disorders or other psychiatric disabilities. Normal physical examination, ecg, laboratorium (blood cells, liver, kidneys)

Ages: 12 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Studypopulation: Patiënts: all female, non -age coupled. Subgroup patients without tube feeding, with tube feeding and a healthy matched control group.
  Control group: healthy volunteers of the University of Maastricht.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
Concentration of ghrelin in blood. | 1 morning

CONTACTS AND LOCATIONS:
Overall Officials: Martine F Delfos, Dr, Principal Investigator — PICOWO Utrecht
Locations (1):
- University Hospital Maastricht, Maastricht, Limburg, Netherlands

REFERENCES:
- [Background] Bosse, T.; Delfos., M.F.; Jonker, C.M. & Treur, J. (2003). Reasoning about adaptive Dynamical Systems in the Analysis of eating Regulation Disorders. N.J. Mahwah. Proceedings of the 25th Annual Conference of the Cognitive Science Society. Lawrence Erlbaum Associates Inc.
- [Background] Both, F. & Delfos, M.F. (in preparation). The role of ghrelin in eating disorders, a review.